CLINICAL TRIAL: NCT01595139
Title: MicroRNAs as Disease Markers for Central Nervous System Tumors in Patients With Neurofibromatosis Type 1
Brief Title: MicroRNAs in Patients With Neurofibromatosis Type 1
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-14927
Record Dates: First submitted 2012-05-08; First posted 2012-05-09 (Estimated); Last update posted 2024-12-06 (Actual); Status verified 2017-07

CONDITIONS: Glioma; Neurofibromatosis Type 1
MeSH Terms: conditions — Glioma; Neurofibromatosis 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NF-1 without evidence of glioma
- NF-1 with evidence of glioma

SUMMARY:
MicroRNAs are small molecules which have recently been discovered in cells. They are known to be responsible for the normal development of cells and when they are disrupted can contribute to the development of cancer. Many previous studies have been done evaluating the expression of microRNAs in normal tissues as well as in a wide variety of cancers.

Recently, microRNAs from tumor cells have been detected circulating in the blood of patients with cancer. This presents a novel opportunity to assess the utility of microRNAs in the blood as an early predictor of cancer as well as a marker of response to therapy. No previous studies have been performed evaluating microRNAs in archived tumor tissue and blood of patients with Neurofibromatosis type 1 (NF-1). The investigators propose a feasibility study to evaluate the presence of microRNAs in archived tumor tissue and the blood of patients with NF-1. If the investigators are able to identify circulating microRNAs in this population of pediatric patients, they will build upon this data in proposing a future study.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 2 years to 21 years.
* Patients with NF-1 being followed in the Neurofibromatosis Clinic.
* Patients have had MRI imaging in the 24 months prior to enrollment on the study.
* Patients may have known concurrent malignancies such as plexiform neurofibroma.
* Patients and/or parents/legal guardians must have signed an informed consent and assent when applicable.

Exclusion Criteria:

* Patients who have had prior tumor-directed therapy (including chemotherapy and/or radiation)
* Patients with a prior or current diagnosis of a malignant peripheral nerve sheath tumor.
* Patients who are considered too ill to participate as determined by their treating physician
* Patients who are pregnant or lactating

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participation in the study will be offered to patient's ages 2 years to 21 years seen for a routine visit in the Neurofibromatosis Clinic at Children's Memorial Hospital and Lurie Children's Hospital in Chicago.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2012-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Evaluate miRNA expression patterns in tissue of low grade gliomas | 2 years

SECONDARY OUTCOMES:
Evaluated miRNA expression patterns between patients with and without imaging findings of gliomas | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Rishi Lulla, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fernandez-L A, Northcott PA, Taylor MD, Kenney AM. Normal and oncogenic roles for microRNAs in the developing brain. Cell Cycle. 2009 Dec 15;8(24):4049-54. doi: 10.4161/cc.8.24.10243. Epub 2009 Dec 5. PMID 19901543
- [Background] Taylor DD, Gercel-Taylor C. MicroRNA signatures of tumor-derived exosomes as diagnostic biomarkers of ovarian cancer. Gynecol Oncol. 2008 Jul;110(1):13-21. doi: 10.1016/j.ygyno.2008.04.033. PMID 18589210
- [Background] Lawrie CH, Gal S, Dunlop HM, Pushkaran B, Liggins AP, Pulford K, Banham AH, Pezzella F, Boultwood J, Wainscoat JS, Hatton CS, Harris AL. Detection of elevated levels of tumour-associated microRNAs in serum of patients with diffuse large B-cell lymphoma. Br J Haematol. 2008 May;141(5):672-5. doi: 10.1111/j.1365-2141.2008.07077.x. Epub 2008 Mar 3. PMID 18318758
- [Background] Mitchell PS, Parkin RK, Kroh EM, Fritz BR, Wyman SK, Pogosova-Agadjanyan EL, Peterson A, Noteboom J, O'Briant KC, Allen A, Lin DW, Urban N, Drescher CW, Knudsen BS, Stirewalt DL, Gentleman R, Vessella RL, Nelson PS, Martin DB, Tewari M. Circulating microRNAs as stable blood-based markers for cancer detection. Proc Natl Acad Sci U S A. 2008 Jul 29;105(30):10513-8. doi: 10.1073/pnas.0804549105. Epub 2008 Jul 28. PMID 18663219
- [Background] Huang Z, Huang D, Ni S, Peng Z, Sheng W, Du X. Plasma microRNAs are promising novel biomarkers for early detection of colorectal cancer. Int J Cancer. 2010 Jul 1;127(1):118-26. doi: 10.1002/ijc.25007. PMID 19876917
- [Background] Ng EK, Chong WW, Jin H, Lam EK, Shin VY, Yu J, Poon TC, Ng SS, Sung JJ. Differential expression of microRNAs in plasma of patients with colorectal cancer: a potential marker for colorectal cancer screening. Gut. 2009 Oct;58(10):1375-81. doi: 10.1136/gut.2008.167817. Epub 2009 Feb 6. PMID 19201770
- [Background] Heneghan HM, Miller N, Lowery AJ, Sweeney KJ, Kerin MJ. MicroRNAs as Novel Biomarkers for Breast Cancer. J Oncol. 2009;2009:950201. doi: 10.1155/2010/950201. Epub 2009 Jul 20. PMID 19639033
- [Background] Zhu W, Qin W, Atasoy U, Sauter ER. Circulating microRNAs in breast cancer and healthy subjects. BMC Res Notes. 2009 May 19;2:89. doi: 10.1186/1756-0500-2-89. PMID 19454029
- [Background] Albers AC, Gutmann DH. Gliomas in patients with neurofibromatosis type 1. Expert Rev Neurother. 2009 Apr;9(4):535-9. doi: 10.1586/ern.09.4. PMID 19344304
- [Background] Chai G, Liu N, Ma J, Li H, Oblinger JL, Prahalad AK, Gong M, Chang LS, Wallace M, Muir D, Guha A, Phipps RJ, Hock JM, Yu X. MicroRNA-10b regulates tumorigenesis in neurofibromatosis type 1. Cancer Sci. 2010 Sep;101(9):1997-2004. doi: 10.1111/j.1349-7006.2010.01616.x. PMID 20550523
- [Background] Smyth GK. Linear models and empirical bayes methods for assessing differential expression in microarray experiments. Stat Appl Genet Mol Biol. 2004;3:Article3. doi: 10.2202/1544-6115.1027. Epub 2004 Feb 12. PMID 16646809
- [Background] J.D. Storey, A direct approach to false discovery rates. JRSS B 64 (2002) 479-498.